CLINICAL TRIAL: NCT06827327
Title: A Randomized Controlled Trial Evaluating the Efficacy of Lactococcus Lactis JCM 5805 (LC-Plasma) Lactic Acid Bacteria in Preventing Upper Respiratory Tract Infections and Reducing Symptom Severity and Duration
Brief Title: LC-Plasma for Preventing URTIs and Reducing Symptoms
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Collaborators: Kirin Holdings Company, Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KURTIS
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-02

CONDITIONS: Healthy Volunteer; URTI
Keywords: LC-Plasma; URTI; Healthy volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LC-Plasma (Experimental): 1 tablet containing 50mg LC-Plasma is taken daily for 24 weeks.
  Interventions: Dietary Supplement: LC-Plasma
- Placebo (Placebo Comparator): 1 tablet containing 50mg microcrystalline cellulose is taken daily for 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: LC-Plasma — 1 tablet containing 50mg LC-Plasma is taken daily for 24 weeks
  Arms: LC-Plasma
Other: Placebo — 1 tablet containing 50mg MCC is taken daily for 24 weeks
  Arms: Placebo

SUMMARY:
The goal of this study is to evaluate the efficacy of the LC-Plasma in preventing upper respiratory tract infections (URTIs) in healthy volunteers. Researchers will compare LC-Plasma to placebo to see if LC-Plasma prevents URTIs. Participants will take a tablet containing LC-Plasma or placebo daily for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-60 years living in Australia
* Individuals with a history of recurrent upper respiratory tract infections
* Able to provide informed consent
* Generally healthy
* Agree to not participate in another clinical trial while enrolled in this trial
* Agree to maintain their usual daily activities without significant changes. This includes not changing their current diet or stopping/starting a new exercise regimen during entire study period
* Agree not to travel internationally for over 1 month in a single trip during the intervention period (baseline to study completion).
* Females of childbearing potential must a prescribed form of birth control

Exclusion Criteria:

* Serious illness e.g., liver disease, kidney disease, heart disease, mood disorders, neurological disorders such as multiple sclerosis.
* Unstable illness e.g., changing medication/treatment.
* BMI <18.5, >30
* Current malignancy (excluding Basal Cell Carcinoma) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years.
* Individuals with chronic respiratory conditions (e.g., asthma, chronic obstructive pulmonary disease).
* Has current symptoms of an acute sickness.
* Active smokers, nicotine use or drug (prescription or illegal substances) abuse
* Current alcohol use (>14 alcoholic drinks week)
* Allergic to any of the ingredients in the active or placebo formula
* Pregnant or lactating woman
* People medically prescribed medications within the last month that would affect the immune and/or the inflammatory response excluding topical steroid use.
* Participants who are currently participating in any other clinical trial or who have participated in any other clinical trial during the past 1 month
* Participants with cognitive damage
* Participants with seasonal allergic rhinitis
* Regular use of antihistamines
* Individuals deemed unsuitable for participation by the Principal Investigator (PI) of this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 650 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence number of URTIs | Day 1 to 24 weeks
  Cumulative incidence number of Upper Respiratory Tract Infections (URTIs)

SECONDARY OUTCOMES:
Cumulative number of infected participants | Day 1 to week 24
  Cumulative number of infected participants
Cumulative number of days that participant recorded symptom positive to WURSS-24 system | Day 1 to week 24
  Cumulative number of days that participant recorded symptom positive to WURSS-24 (Wisconsin Upper Respiratory Symptom Survey) scoring system during intervention period.
Cumulative scores of each parameter in WURSS-24 scoring system, as well as the total sum of all parameters for each participant. | Day 1 to week 24
  Cumulative scores of each parameter in WURSS-24 scoring system during the intervention period, as well as the total sum of all parameters for each participant.
Length of URTI symptomatic days per one URTI episode. | Day 1 to week 24
  Length of Upper Respiratory Tract Infection (URTI) symptomatic days per one URTI episode.

OTHER OUTCOMES:
Safety: Occurrence of adverse events and Serious Adverse Events | Day 1 to week 24
  Occurrence of adverse events and Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Yusuke Ushida, Study Director — Kirin Holdings Company, Limited; Osamu Kanauchi, Study Director — Kirin Holdings Company, Limited
Locations (1):
- RDC Clinical, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No